CLINICAL TRIAL: NCT06938659
Title: Comparison of Low Dose Emicizumab and Low Dose Factor VIII as a Prophylaxis in Hemophilia A Patients- a Randomized Control Trial'
Brief Title: Low Dose Emicizumab vs Low Dose Factor VIII in Prophylaxis in Hemophilia A Patients
Acronym: AFEEL
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Akhil Ranjon Biswas, Professor and Head of the Department of Hematology., Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2024/215
Record Dates: First submitted 2025-03-12; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia A
Keywords: Low dose Factor VIII; Low dose Emicizumab; Prophylaxis; Hemophilia A with inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab; Factor VIII; F8 protein, human

STUDY DESIGN:
Intervention Model Description: we will select 20 severe hemophilia A patients randomly from interested patients. we will randomize 6 patients with inhibitor to factor VIII in Low dose Emicizumab with Inhibitor group (I) and rest 14 will be randomized by block randomization in Low dose Emicizumab (without inhibitor-WI) and low dose Factor VIII group.
  patients with inhibitor (Emicizumab Group-I):
  Patients without inhibitor (Emicizumab Group-WI):
  Patients without inhibitor (Factor VIII Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Emicizumab Group- I (Experimental): Severe hemophilia A patients with inhibitor
  Interventions: Drug: Emicizumab Injection
- Emicizumab Group- WI (Experimental): Severe hemophilia A Patients without inhibitor (Emicizumab Group):
  Interventions: Drug: Emicizumab Injection
- Factor VIII Group (Active Comparator): Severe hemophilia A Patients without inhibitor.
  Interventions: Drug: Factor VIII (FVIII)

INTERVENTIONS:
Drug: Emicizumab Injection — Emicizumab 0.8-1.5mg/kg weekly for 4 weeks as loading dose. Then 0.8-1.5mg/kg 4-weekly for 24 weeks will be used in Emicizumab group-I and Emicizumab Group- WI
  Other Names: Hemlibra
  Arms: Emicizumab Group- I; Emicizumab Group- WI
Drug: Factor VIII (FVIII) — 10-15 unit/Kg thrice weekly (for conventional half-life products) or twice weekly (for extended half-life products) for 28 weeks. Inj. Factor VIII is available in 250U, 500U, 750U & 1,000 IU vail sizes. Dose will be round up to full nearest full vail strength.
  Other Names: Afstyla; Kovaltry
  Arms: Factor VIII Group

SUMMARY:
Low dose factor VIII prophylaxis is practiced around the world. Role of standard dose Emicizumab prophylaxis is well established. Emicizumab is an expensive drug. Standard dose Emicizumab prophylaxis is very expensive for hemophilia A patients and troublesome for government to ensure continuous supply. This study intends to compare low dose Factor VIII prophylaxis with low dose Emicizumab prophylaxis and compare whether low dose Emicizumab is as effective as low dose Factor VIII prophylaxis. So, it is possible to continue prophylaxis program in hemophilia A patients with a cost-effective way in our country without risking the patient health. Moreover, Emicizumab prophylaxis reduces the chance of developing inhibitor to Factor VIII and it is convenient for administration due to less frequent and subcutaneous administration. 20 severe hemophilia A patients will be selected randomly from interested patients for this study. 6 patients with inhibitor will be randomized in Low dose Emicizumab with Inhibitor group (I) and rest 14 will be randomized by block randomization in Low dose Emicizumab (without inhibitor-WI) and low dose Factor VIII group at 4:10 ratio. Initial loading dose will be given and the participants will be followed up for 6 months. At the end of the study Annualized bleeding rate (ABR), Annualized joint bleeding rate (AJBR), Annualized spontaneous bleeding rate (ASBR), APTT will be compared among the groups. Inhibitor to factor VIII will also be evaluated after six months in Factor VIII group.

DETAILED DESCRIPTION:
Selection criteria for the study- Severe hemophilia A patients with or without inhibitor to factor VIII will be eligible to participate in the study. Patients with inhibitor will not be included in factor VII group.

Sample Size: Sample size is determined by availability of drugs rather than any scientific formula. The investigators can provide Emicizumab to 10 patients for 28 weeks as prophylaxis. So, the investigators intend to include 10 patients in each group.

Sampling technique: The investigators will select 20 severe hemophilia A patients randomly from interested patients. The investigators will randomize 6 patients with inhibitor in Low dose Emicizumab with Inhibitor group (I) and rest 14 will be randomized by block randomization in Low dose Emicizumab (without inhibitor-WI) and low dose Factor VIII group at 4:10 ratio Variables to be studied- A. Independent variable

1. Socio-demographic variables- Age, Educational status, Weight, Occupation
2. Variables related to Hemophilia- Presence of Inhibitor B. Dependent variable

1. Main outcome variables- Annualized bleeding rate (ABR), Annualized joint bleeding rate (AJBR), Annualized spontaneous bleeding rate (ASBR), APTT 2. Confounding variables- Development of new inhibitor to factor VIII Patients and/or parents will be thoroughly informed about the study, drugs to be used, risk & benefits and follow up plan. Their consent for this study will be taken and they will be enrolled in the study. For Participants under 18 years, consent will be obtained from parents or legal guardian. Participants ≥18 years will give his/her own consent. Randomization will be generated by computer.

Dose- Emicizumab 0.8-1.5mg/kg weekly for 4 weeks as loading dose. Then 0.8-1.5mg/kg 4-weekly for 24 weeks. Inj. Emicizumab has 30mg in vail. Dose will be rounded to 30mg, 60 mg or any dose nearest to 1 mg/kg when fractionation of vail is possible.

Factor VIII- 10-15 unit/Kg thrice weekly (for conventional half-life products) or twice weekly (for extended half-life products) for 28 weeks. Inj. Factor VIII is available in 250U, 500U, 750U & 1,000 IU vail sizes. Dose will be round up to full nearest full vail strength.

Follow Up- Participants in Emicizumab group will visit weekly for first 4 week than once in every 4 week for 24 weeks (Total 28 weeks).

Participants in Factor VIII group will visit twice weekly for 28 weeks. Information of data collection sheet will be collected once in a week.

Patient must attend physically for every dose administration. He will be asked for number of bleeding- traumatic, spontaneous bleeding, joint bleeding, frequency of hospital visit due to hemophilia related problems in between doses and investigate for APTT.

Primary End Point- This study will include 28 weeks follow up of the patients. Each patient will receive 28 weeks prophylaxis. After that period patients will continue prophylaxis if drugs are available but will not be considered for this study. Otherwise, they will receive on demand treatment in our HTC (hemophilia treatment center).

Supportive care and rescue- A Data and Safety Monitoring Board (DSMB) will be formed which will include members suggested by IRB. Any adverse event or serious adverse event (will be delt with proper medical care.

If any patient developed spontaneous or traumatic bleeding episode during prophylaxis, they will be treated with standard dose on demand treatment on priority basis.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A patient with or without inhibitor to factor VIII.

Exclusion Criteria:

* 1. Severe hemophilia A patient not willing to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean of Annualized bleeding rate (ABR) among the study groups will be compared. | 06 months
  ABR will be calculated as the number of reported bleeding events divided by 06 (the number of months in the reporting time window) and multiplied by 12. e.g. if a participant total bleeding event are 12 in 6 months, ABR of this patients is 12/6*12=24
Mean of Annualized joint bleeding rate (AJBR) among the study groups will be compared. | 06 months
  AJBR will be calculated as the number of reported joint bleeding events divided by 06 (the number of months in the reporting time window) and multiplied by 12. e.g. if a participant Joint Bleeding event is 6 in 6 months than AJBR will be 6/6*12=12.
Mean of Annualized spontaneous bleeding rate (ASBR) among the study groups will be compared. | 06 months
  ASBR will be calculated as the number of reported spontaneous bleeding events divided by 06 (the number of months in the reporting time window) and multiplied by 12. e.g. if a participant has total 4 spontaneous bleeding event in six months than ASBR will be 4/6*12= 7.99
Mean of APTT among the groups will be compared. | 06 months
  APTT

SECONDARY OUTCOMES:
Inhibitor to Factor VIII- | 06 months
  Check for development of inhibitor to Factor VIII in Factor VIII group and emicizumab group without inhibitor.

CONTACTS AND LOCATIONS:
Overall Officials: Akhil R. Biswas, MBBS, FCPS, Principal Investigator — Dhaka Medical College
Locations (1):
- Dhaka Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Participants annual Bleeding rate, Factor level, inhibitor status, dose of drugs
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 01.06.2025 to 30.05.2030
Access Criteria: We can share information to doctors by e-mail.

REFERENCES:
- [Result] Shima M, Hanabusa H, Taki M, Matsushita T, Sato T, Fukutake K, Kasai R, Yoneyama K, Yoshida H, Nogami K. Long-term safety and efficacy of emicizumab in a phase 1/2 study in patients with hemophilia A with or without inhibitors. Blood Adv. 2017 Sep 27;1(22):1891-1899. doi: 10.1182/bloodadvances.2017006684. eCollection 2017 Oct 10. PMID 29296836
- [Result] Young G, Liesner R, Chang T, Sidonio R, Oldenburg J, Jimenez-Yuste V, Mahlangu J, Kruse-Jarres R, Wang M, Uguen M, Doral MY, Wright LY, Schmitt C, Levy GG, Shima M, Mancuso ME. A multicenter, open-label phase 3 study of emicizumab prophylaxis in children with hemophilia A with inhibitors. Blood. 2019 Dec 12;134(24):2127-2138. doi: 10.1182/blood.2019001869. PMID 31697801
- [Result] Xu Y, Wang Y, Wu R, Zheng C, Zhang L, Xu W, Feng X, Wang H, Cao X, He L, Xue T, Jin M, Xie B, Ling J, Sun L, Su R, Cheng H, Fang Y, Poon MC, Liu W, Zhang L, Xue F, Yang R. Reduced doses of emicizumab achieve good efficacy: Results from a national-wide multicentre real-world study in China. Haemophilia. 2024 Jul;30(4):959-969. doi: 10.1111/hae.15062. Epub 2024 Jun 9. PMID 38853005

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT06938659/Prot_SAP_ICF_000.pdf